CLINICAL TRIAL: NCT02051933
Title: The Effect of Botulinum Toxin A Injections on Ankle Dorsiflexion Following Internal Fixation of Tibial Plafond (Pilon) Fractures: A Pilot Study
Brief Title: The Effect of Botulinum Toxin A Injections on Ankle Dorsiflexion Following Internal Fixation of Tibial Pilon Fractures
Acronym: Botox
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-12-19B
Record Dates: First submitted 2013-10-14; First posted 2014-01-31 (Estimated); Results first posted 2022-02-25 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-02

CONDITIONS: Equinus Contracture
Keywords: pilon; tibial plafond; botox; ankle dorsiflexion; ankle functionality; ankle range of motion
MeSH Terms: conditions — Equinus Deformity | interventions — Botulinum Toxins, Type A; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox (Active Comparator): Botox: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator): Placebo: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL 0.9% sodium chloride solution . The dose of 0.9% sodium chloride will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Placebo will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in placebo(rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Botulinum toxin type A — At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
  Other Names: Botox
  Arms: Botox
Drug: sodium chloride — At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL 0.9% sodium chloride solution . The dose of 0.9% sodium chloride will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Placebo will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in placebo(rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if botulinum toxin type A (Botox) injections, at the time of surgery for pilon fractures, will improve ankle range-of-motion and functionality.

DETAILED DESCRIPTION:
To determine if the use of Botulinum toxin A intramuscular injections of the gastrocsoleus complex in patients with operatively treated tibial plafond fractures will result in:

1. increased ankle dorsiflexion when compared to controls
2. increased ankle functionality as measured by the FAAM, and quality of life as measured by the SF-36, when compared to controls
3. a higher proportion of patients achieving at least 10 degrees of dorsiflexion when compared to controls

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older with a tibial plafond fracture to be treated by a staged protocol involving primary external fixation and definitive fixation within 3 weeks from the injury.

(Non-definitive, interval procedures such as repeat irrigation and debridement and fibular fixation are allowed.)

Exclusion Criteria:

* Younger than 18 years of age
* Significant traumatic brain injury or cognitive disability that would interfere with post-operative rehabilitation and study questionnaires
* Nerve, vascular, or tendon injury of the lower leg: injury to the tibial or peroneal motor nerves, injury to the posterior tibial artery requiring repair, or laceration of tendons that are involved in plantar flexion or dorsiflexion of the ankle which require repair
* History of prior lower extremity fracture to the tibia or ankle of the affected limb.
* Incarcerated patients.
* Patients unable or unwilling to return for follow-up examination.
* Pregnant or lactating patients.
* History of disease affecting the neuromuscular junction (ex: myasthenia gravis).
* Use of aminoglycoside antibiotics at the time of definitive fixation.
* Ipsilateral foot injury that will impair dorsiflexion exercises: Lisfranc injuries, fractures or dislocations of the talus, calcaneus, navicular, cuboid, cuneiforms, or metatarsals (phalanx fractures or dislocations will not be excluded).
* Patients receiving Botulinum Toxin A for other reasons.
* Patients with a known hypersensitivity to Botulinum toxin A.
* Gustilo Anderson type III B and C.
* Patients with a weight greater than 115 kg - to ensure proper injection locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav A Karunakar, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botox | Placebo
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Botulinum Toxin Type A: Botox: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
- 0.9% Sodium Chloride: Placebo: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL 0.9% sodium chloride solution . The dose of 0.9% sodium chloride will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Placebo will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in placebo(rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (8.9) | 42.0 (11.0) | 43.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ankle Dorsiflexion of Injured Extremity
Description: The difference in ankle dorsiflexion between the injured and un-injured ankles as measured with goniometer 6 month from surgery.
Time Frame: 6 month follow-up visit
Measure: Mean (Full Range); unit: degrees
Groups:
- Botox: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 4 | 4
degrees | -3.8 [-12 to 5] | 11.8 [-3 to 40]

2. Secondary Outcome: Short Form-36 (SF-36)Health Related Quality of Life
Description: The SF-36 is a patient reported survey of health. Physical functioning, role functioning/physical and general health sub-scores ranges from 0 (worst)- 100 (best)
Time Frame: 6 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botox: See Botox intervention description:
  Botox: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
- Placebo: See Placebo Intervention Description
  Placebo: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL 0.9% sodium chloride solution . The dose of 0.9% sodium chloride will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Placebo will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in placebo(rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  SF-36 Physical Functioning) | 30.0 (24.5) | 55.0 (16.8)
  SF-36 Role functioning/physical | 0 (0) | 0 (0)
  SF-36 General health | 65.0 (21.6) | 68.8 (18.9)

3. Secondary Outcome: Short Form-36 (SF-36) Health Related Quality of Life
Description: as for outcome 2
Time Frame: 12 month follow-up visits
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botox: See Botox intervention description:
  At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale
  SF-36 Physical Functioning) | 45.0 (36.1) | 70.0 (13.2)
  SF-36 Role functioning/physical | 58.3 (52.0) | 33.3 (38.2)
  SF-36 General health | 63.3 (37.5) | 75.0 (26.5)

4. Secondary Outcome: Ankle Pain at 6 Month
Description: Brief pain inventory (BPI) severity subscale measures pain severity with a higher score indicates worse pain (10) and lower score of no pain (0). The pain interference subscale of the BPI measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Time Frame: 6 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botox: Botulinum toxin A solution
  Botulinum toxin A: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL Botulinum toxin type A. The dose of botulinum toxin will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Botox will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in Botox (rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
- Placebo: 0.9% sodium chloride solution
  Placebo: At the time of definitive fixation, the hospital's investigational pharmacy will provide four syringes containing 0.5mL 0.9% sodium chloride solution . The dose of 0.9% sodium chloride will be calculated based on the patient's weight in kilograms, such that a total dose of 200U of Placebo will be used for a 70kg individual. The dosage will scale linearly in proportion to the patient's body weight, such that each kilogram change results in a 3U change in placebo(rounded to the nearest 30U interval change from 200U, with a maximum of 300U).
  45-55 kg: 140U 55-65 kg: 170U 65-75 kg: 200U 75-85 kg: 230U 85-95 kg: 260U 95-105 kg: 290U 105-115 kg: 300U
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  Pain Severity (BPI) | 3.38 (1.9) | 2.94 (1.2)
  Pain Interference (BPI) | 3.4 (2.4) | 1.7 (2.6)

5. Secondary Outcome: Ankle Pain at 12 Month
Description: as for outcome 4
Time Frame: 12 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale
  Pain Severity (BPI) | 2.92 (2.5) | 3.17 (1.4)
  Pain Interference (BPI) | 4.1 (3.5) | 1.0 (1.0)

6. Secondary Outcome: Functional Status of the Ankle at 6 Month
Description: The Foot and Ankle Ability Measure (FAAM) will be obtained to assess the functional status of the affected ankle.
  Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Item score totals, which range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were transformed to percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction.
Time Frame: 6 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 32.4 (19.0) | 65.2 (20.7)

7. Secondary Outcome: Functional Status of the Ankle at 12 Month
Description: The Foot and Ankle Ability Measure (FAAM) will be obtained to assess the functional status of the affected ankle. A higher score represents a higher level of physical function.
Time Frame: 12 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 63.1 (12.5) | 70.2 (16.9)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Botox | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-09-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT02051933/Prot_SAP_000.pdf
  • Informed Consent Form (2013-04-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02051933/ICF_001.pdf